CLINICAL TRIAL: NCT06029140
Title: Stereotactic Radiotherapy Management of Brain Metastases: the Value of a Longitudinal Multimodal Approach
Brief Title: Stereotactic Radiotherapy Management of Brain Metastases: the Value of a Longitudinal Multimodal Approach (POSTPONE)
Acronym: POSTPONE
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: University Hospital, Brest (Other)
Responsible Party: Sponsor
Other Study IDs: 29BRC23.0143 - POSTPONE
Record Dates: First submitted 2023-08-01; First posted 2023-09-08 (Actual); Last update posted 2024-08-09 (Actual); Status verified 2023-09

CONDITIONS: Brain Metastases, Adult
Keywords: stereotactic radiotherapy; radionecrosis; local relapse; PET DOPA; Multimodal MRI
MeSH Terms: conditions — Brain Neoplasms

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
The management of brain metastases has evolved́ rapidly in recent years. It is estimated that 20% to 40% of cancer patients will develop brain metastases (BM) during the course of their disease. Whole-brain radiotherapy has long been the first-line treatment for brain metastases. However, large-scale international clinical trials conducted over the past decade have established stereotactic radiotherapy (SR) as the treatment of choice for the management of brain metastases (BM). However, even though the method of radiation delivery has evolved considerably, the problem of monitoring and managing brain metastases remains unresolved.

This study therefore has several focuses:

1. Evaluation of the benefit of early remnographic assessment (6 weeks): impact on recurrence-free survival and overall survival.
2. Evaluation of a diagnostic approach to radionecrosis: complementarity of DOPA PET and multimodal MRI.
3. The benefits of longitudinal remnographic monitoring with the development of segmentation and automated follow-up tools

DETAILED DESCRIPTION:
The management of brain metastases has evolved́ rapidly in recent years. It is estimated that 20% to 40% of cancer patients will develop brain metastases (BM) during the course of their disease. Whole-brain radiotherapy has long been the first-line treatment for brain metastases. However, large-scale international clinical trials conducted over the past decade have established stereotactic radiotherapy (SRT) as the treatment of choice for the management of brain metastases (BM). However, even though the method of radiation delivery has evolved considerably, the problem of monitoring and managing brain metastases remains unresolved. Indeed, BM patients constitute a growing population due to the increased efficacy of systemic treatments, making the occurrence of BM higher. Management of the disease is not only aimed at alleviating symptoms and, initially, improving survival, but must also take into account patients' quality of life. Patients with a poor prognosis should not be over-treated, while those with a more favorable prognosis should not be under-treated.

With this in mind, a number of tools were rapidly developed to grade the prognosis of patients with BM. Recursive partitioning analysis (RPA) and Graded Prognostic Assessment (GPA) are the main ones. They are based on prognostic factors that include age, Karnofsky index, primary tumor control, presence of extracerebral localization, histological type and presence of genetic mutations for each primary. Finally, we must also take into account the growing involvement of systemic treatments in the control of brain disease when the blood-brain barrier (BBB) is crossed.

Several studies have shown that patients with symptomatic cerebral recurrences have poorer survival and generate higher costs for the healthcare system than asymptomatic patients whose recurrences have been detected by routine surveillance imaging. The importance of frequent surveillance imaging is therefore essential. National Comprehensive Cancer Network (NCCN) recommendations include MRI every 2-3 months for the first year, then every 4-6 months indefinitely. The recommendations of the Association des Neuro-Oncologues d'Expression Française (ANOCEF) recommend brain MRI at least every 3 months for the first year (9), RECORAD recommends MRI surveillance every 3 months for the first 2 years, then every 6 months (10), and Cancer Care Ontario Organization (CCO) recommends a 1st follow-up MRI 2 to 3 months after the end of treatment, followed by MRI surveillance every 2 to 3 months for 1 year, and MRI surveillance every 3 to 4 months for 2 to 3 years. Given the heterogeneity of follow-up modalities, and the absence of any recommendation for surveillance MRI imaging earlier than 3 months after treatment, the Brest University Hospital decided to carry out an early remnographic reassessment of patients treated with intracerebral stereotactic radiotherapy 6 weeks after the end of treatment, and then every 3 months for a minimum of 2 years.

After SRT for brain metastases, the median time to development of a radiation-induced adverse event or radionecrosis is 7 to 11 months. Similarly, the risk of local tumor recurrence after SR is < 5% after 18 months. In terms of complications, improvements in systemic therapy mean that patients are living longer and are at greater risk of tumour recurrence later than previously (defined as > 18 months after SRT). Radionecrosis may therefore occur in up to 50% of patients several months to several years after irradiation, depending on several factors, including dose fractionation patterns and the volume of normal brain receiving high-dose irradiation.

Radionecrosis can produce symptoms difficult to distinguish from those of local progression and, if left untreated, can lead to significant morbidity and mortality. Correct differential diagnosis between radionecrosis and local progression is extremely important, as the two situations must be managed differently. Surgery or re-irradiation is generally proposed as salvage therapy in patients with local progression, whereas radionecrosis is most often treated with corticosteroids.

Differential diagnosis between radiation-induced changes and brain tumor recurrence is a challenge in the treatment of brain metastases. The RANO (Response Assessment in Neuro-Oncology) group has recognized that an approach based on a single imaging modality is insufficient to establish a correct diagnosis. It recommends the use of advanced imaging techniques, such as MRI with diffusion sequence and perfusion map, spectroscopy and PET.

Several radiopharmaceuticals, including the amino acid tracers O-(2-[18F]fluoroethyl)-L-tyrosine (FET) and 3,4-dihydroxy-6-[18F]-fluoro- l-phenylalanine (F-DOPA), have proved useful in distinguishing radionecrosis from local progression in patients with brain metastases.

Several observations can therefore be made:

* Heterogeneity of practices concerning remnographic surveillance, particularly at an early stage.
* Heterogeneity in practices concerning suspicion of radionecrosis

This study therefore has several focuses:

1. Evaluation of the benefit of early remnographic assessment (6 weeks): impact on recurrence-free survival and overall survival.
2. Evaluation of a diagnostic approach to radionecrosis: complementarity of DOPA PET and multimodal MRI.
3. The benefits of longitudinal remnographic monitoring with the development of segmentation and automated follow-up tools

ELIGIBILITY:
Inclusion Criteria:

* Age ≥ 18 years
* Patients with solid cancer with brain metastases treated by hypofractionated external stereotactic radiotherapy at the CHRU de Brest between 01/01/2014 and 31/12/2022
* Patient affiliated to a social security scheme

Exclusion Criteria:

* Patients with primary brain tumors
* Patients treated with normofractionated external cerebral radiotherapy
* Age < 18 years
* Patients under legal protection (guardianship, curatorship, etc.)

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patient treated with intracerebral stereotactic radiotherapy at the Brest University Hospital as part of the management of a secondary localization of a primary solid cancer.
Sampling Method: Non-Probability Sample
Enrollment: 700 (Estimated)
Dates: Start 2023-08-01 (Actual); Primary Completion 2024-07-01 (Actual); Study Completion 2024-09-01 (Estimated)

PRIMARY OUTCOMES:
Risk factors of radionecrosis | Through study completion, an average of 1 year
  The main objective is to identify risk factors for cerebral radionecrosis after stereotactic radiotherapy in patients treated for brain metastases.

SECONDARY OUTCOMES:
Risk factors of local relapse | Through study completion, an average of 1 year
  Clinical, dosimetric and radiological factors influencing local control
Post-SRT follow-up | Through study completion, an average of 1 year
  Practical analysis of the benefits of performing MRI 6 weeks after the end of stereotactic radiotherapy treatment, and determining precise criteria to better target patients who would benefit most from it.

OTHER OUTCOMES:
Automatic segmentation of brain metastasis | Through study completion, an average of 1 year
  Development of a deep-learning algorithm for the automatic segmentation on MRI, CT and CT scanners
Automatic follow-up | Through study completion, an average of 1 year
  Development of a deep-learning algorithm for the automatic longitudinal follow-up

CONTACTS AND LOCATIONS:
Overall Officials: Vincent Bourbonne, MD, PhD, Principal Investigator — Radiation Oncology Department, Brest University Hospital
Locations (1):
- Chu Brest, Brest, France

IPD SHARING:
Plan to Share IPD: Yes
All collected data that underlie results in a publication
Supporting Information: Study Protocol
Time Frame: Data will be available beginning three years and ending fifteen years following the final study report completion
Access Criteria: Data access requests will be reviewed by the internal committee of Brest UH. Requestors will be required to sign and complete a data access agreement